CLINICAL TRIAL: NCT07274787
Title: An Open Label, Prospective, Pilot Study To Evaluate The Safety And Effectiveness Of The NaviFUS System In Conjunction With A Standard Treatment Regimen Of Bevacizumab (BEV) In Patients With Recurrent Glioblastoma
Brief Title: Safety And Effectiveness Of NaviFUS System With Bevacizumab In Recurrent Glioblastoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: NaviFUS Corporation (Industry)
Responsible Party: Principal Investigator, Kyle Wang, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-BN-24-01
Record Dates: First submitted 2025-11-20; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: GBM
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NaviFUS + bevacizumab (Experimental): NaviFUS system with concomitant microbubble administration in conjunction with bevacizumab (BEV)
  Interventions: Device: NaviFUS System; Drug: Lumason; Drug: Bevacizumab

INTERVENTIONS:
Device: NaviFUS System — The NaviFUS System is a FUS phased array system intended to transcranially deliver burst-mode ultrasound energy with the concurrent microbubble intravenous administration to temporally and locally open the BBB. The NaviFUS System is indicated for use to enhance the permeability of conventionally administered therapeutic agents into targeted brain tissue to enhance their therapeutic effects.
Drug: Lumason — The NaviFUS System is a FUS phased array system intended to transcranially deliver burst-mode ultrasound energy with the concurrent microbubble intravenous administration to temporally and locally open the BBB.
Drug: Bevacizumab — In this proposed clinical investigation, the NaviFUS System will be used in conjunction with BEV in recurrent GBM patients.

SUMMARY:
This study will evaluate the safety and early effectiveness of the NaviFUS system with concomitant microbubble administration in conjunction with BEV in recurrent GBM patients.

DETAILED DESCRIPTION:
The primary objective of this clinical investigation is to evaluate the safety of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.

Safety will be assessed using the following methods: Device-related Adverse Events (AEs) reported [Time Frame: Through study completion, up to 24 weeks].

To determine the incidence and severity of device-related AEs for bevacizumab plus NaviFUS System treatment in patients with recurrent glioblastoma multiforme (rGBM), the following safety parameters will be assessed: AEs, physical examination (PE), vital signs, neurological examination (NE), Karnofsky Performance Status (KPS), Mini-Mental State Examination (MMSE), clinical laboratory tests, proteinuria, and ECG.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female patients ≥ 18 years of age.
2. Histologically confirmed glioblastoma at original diagnosis, recurrent after prior radiotherapy and temozolomide chemotherapy.
3. Must have measurable disease ≥ 10mm (according to RANO criteria) .
4. Interval since completion of radiation treatment (including radiation at original diagnosis and/or radiation for recurrent disease) ≥ 12 weeks.
5. If on steroids, must be on a stable dose for ≥ 7 days prior to study treatment.
6. Body mass index (BMI) ≥17 kg / m2.
7. Minimum interval since last drug therapy:

   1. 1 week for non-cytotoxic agents (e.g., interferon, tamoxifen), daily chemotherapy (e.g., metronomic temozolomide, cytoxan) or targeted therapies administered daily (e.g., gleevec, tarceva).
   2. 4 weeks since last cytotoxic therapy.
   3. 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen (e.g., carmustine).
8. Life expectancy ≥ 12 weeks.
9. KPS Score > 60.
10. Adequate hepatic, renal, coagulation, and hematopoietic function:

    1. Hemoglobin ≥ 8 g/dL.
    2. Platelets ≥ 100,000/mm3.
    3. Neutrophils ≥ 1,500/mm3.
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN).
    5. Urine protein creatinine (UPC) ratio < 1 or urine dipstick for proteinuria ≤ 2+.
    6. Alanine transaminase (ALT) < 3 x ULN.
    7. Aspartate transaminase (AST) < 3 x ULN.
    8. Prothrombin time ≤ 1.2 x ULN.
    9. International Normalized Ratio (INR) < 1.5.
    10. Bilirubin < 2 x ULN.
11. Center of region of interest (ROI) (i.e., tumor site) ≥30mm deep to skull bone.
12. If there is the potential for pregnancy, must agree to follow acceptable birth control methods to avoid conception.
13. Able and willing to have their hair shaved (either whole head or the region where the coupling membrane will touch) and placement of peripheral IV line prior to treatment.

Exclusion Criteria:

* 1) Previous treatment with an inhibitor of vascular endothelial growth factor (VEGF) or VEGF receptor (VEGFR), including bevacizumab.

  2) New York Heart Association (NYHA) Grade II or greater congestive heart failure requiring hospitalization within 12 months prior to screening.

  3) Hypertension (systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 100 mmHg).

  4) Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, severe cerebral or myocardial infarction, cardiac shunt, heart attack within the previous 12 months, stroke (except for transient ischemic attack; TIA) within the previous 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.

  5) Unstable Pulmonary Disease or Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of screening.

  6) Implanted pacemaker, defibrillator or deep brain stimulator, or other implanted electronic devices in the brain or documented clinically significant arrhythmias.

  7) Major surgery such as intra-thoracic, intra-abdominal or intra-pelvic (with the exception of craniotomy), open biopsy or significant traumatic injury ≤ 4 weeks prior to screening, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to screening, or who have not recovered from side effects of such procedure or injury.

  8) Known human immunodeficiency virus (HIV) positivity.

  9) Acute bacterial or fungal infection requiring intravenous antibiotics at the time of screening.

  10) Pregnant or breast-feeding women.

  11) Known sensitivity/allergy to MRI contrast agents, CT contrast agents, SonoVue® [Lumason®], bevacizumab, or any of their components.

  12) Abnormal baseline findings considered by the Investigator to indicate conditions that might affect study endpoints.

  13) Hemorrhage or cyst within the ROI.

  14) ROI in the deep center brain with crucial brain functions, such as in the region of the brain stem.

  15) The receipt of an investigational drug within a period of 4 weeks prior to the first FUS exposure.

  16) Use of any recreational drugs or a history of drug addiction.

  17) Difficulty lying supine and still for the FUS procedure length.

  18) Any other condition that, in the Investigator's judgment, might increase the risk to the patient or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety -assessed using -Device-related Adverse Events (AEs) reported | Through study completion, up to 24 weeks
  The primary objective of this clinical investigation is to evaluate the safety of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  Safety will be assessed using the following methods: Device-related Adverse Events (AEs) reported [Time Frame: Through study completion, up to 24 weeks].

SECONDARY OUTCOMES:
Progression-free survival at 6-months and 12-months as determined using the Radiologic Assessment in Neuro-Oncology (RANO) criteria. | Pr6-months and 12-months
  The secondary objective of this clinical investigation is to evaluate the effectiveness of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  1) Progression-free survival at 6-months and 12-months as determined using the Radiologic Assessment in Neuro-Oncology (RANO) criteria.
Median PFS at 6-months and 12-months as determined using the RANO criteria | 6-months and 12-months
  The secondary objective of this clinical investigation is to evaluate the effectiveness of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  2) Median PFS at 6-months and 12-months as determined using the RANO criteria
Objective response rate (ORR) as determined using the RANO criteria at Week 8, 16, and 24. | Week 8, 16, and 24.
  The secondary objective of this clinical investigation is to evaluate the effectiveness of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  3) Objective response rate (ORR) as determined using the RANO criteria at Week 8, 16, and 24.
Overall survival (OS) at 6 & 12 months. | 6 & 12 months
  The secondary objective of this clinical investigation is to evaluate the effectiveness of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  4) Overall survival (OS) at 6 & 12 months.
Median OS at 18 months. | 18 months.
  The secondary objective of this clinical investigation is to evaluate the effectiveness of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  5) Median OS at 18 months.
Change in contrast enhancement (intensity) in MRI following BBB disruption at Week 8, 16, and 24 compared to baseline (Week 0). | Week 8, 16, and 24 compared to baseline (Week 0).
  The secondary objective of this clinical investigation is to evaluate the effectiveness of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  6) Change in contrast enhancement (intensity) in MRI following BBB disruption at Week 8, 16, and 24 compared to baseline (Week 0).
Change in corticosteroid use at Week 2, 4, 6, and 8 compared to baseline (Week 0). | Week 2, 4, 6, and 8 compared to baseline (Week 0).
  The secondary objective of this clinical investigation is to evaluate the effectiveness of BEV combined with the NaviFUS System for the treatment of patients with recurrent GBM.
  7) Change in corticosteroid use at Week 2, 4, 6, and 8 compared to baseline (Week 0).
Change in quality of life (QoL) as determined by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) at Week 4, 8, and 16 compared to baseline (Week 0). | Week 4, 8, and 16 compared to baseline (Week 0).
  Change in quality of life (QoL) as determined by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) at Week 4, 8, and 16 compared to baseline (Week 0).
  1. Lower scores indicate better QoL out comes whereas higher scores indicate a poorer OoL outcomes.
  2. Minimum score is 0, Maximum score is: 112
Change in quality of life (QoL) as determined by the Brain Cancer Questionnaire (BN20) at Week 4, 8, and 16 compared to baseline (Week 0). | Week 4, 8, and 16 compared to baseline (Week 0).
  Change in quality of life (QoL) as determined by the Brain Cancer Questionnaire (BN20) at Week 4, 8, and 16 compared to baseline (Week 0).
  1. Lower scores indicate better QoL out comes whereas higher scores indicate a poorer OoL outcomes.
  2. Minimum score is 0, Maximum score is: 112

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided